CLINICAL TRIAL: NCT04428151
Title: A Phase 2, Randomized, Open-label Three-arm Clinical Study to Evaluate the Safety and Efficacy of Lenvatinib (E7080/MK-7902) in Combination With Pembrolizumab (MK-3475) Versus Standard of Care Chemotherapy and Lenvatinib Monotherapy in Participants With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC) That Have Progressed After Platinum Therapy and Immunotherapy (PD-1/PD-L1 Inhibitors) (LEAP-009)
Brief Title: Lenvatinib (E7080/MK-7902) in Combination With Pembrolizumab (MK-3475) vs. Standard Chemotherapy and Lenvatinib Monotherapy in Participants With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma That Progressed After Platinum Therapy and Immunotherapy (MK-7902-009/E7080-G000-228/LEAP-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7902-009; LEAP-009 (Other: MSD); E7080-G000-228 (Other: Eisai); MK-7902-009 (Other: MSD); 2022-500820-31-00 (Registry Identifier: EU CT); U1111-1278-2707 (Registry Identifier: UTN); 2019-000569-19 (EudraCT Number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — lenvatinib; pembrolizumab; Docetaxel; Capecitabine; Paclitaxel; Cetuximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lenvatinib + Pembrolizumab (Experimental): Participants will be treated with the combination of lenvatinib (once daily 20 mg oral dose) plus pembrolizumab (200 mg 30-minute intravenous (IV) infusion on Day 1 of each 21-day cycle for 35 cycles), until centrally verified disease progression, or until a protocol-specified discontinuation criterion is met. Participants may receive up to an additional 17 cycles of pembrolizumab as Second Course treatment, with or without lenvatinib.
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab
- SOC Chemotherapy (Active Comparator): Participants will be treated with investigator's choice of standard of care (SOC) chemotherapy (docetaxel, paclitaxel, cetuximab, or capecitabine) until centrally verified disease progression, or until a protocol-specified discontinuation criterion is met.
  Interventions: Drug: Docetaxel; Drug: Capecitabine; Drug: Paclitaxel; Drug: Cetuximab
- Lenvatinib Monotherapy (Active Comparator): Participants will be treated with lenvatinib monotherapy (once daily 24 mg oral dose) until centrally verified disease progression, or until a protocol-specified discontinuation criterion is met.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — 20 mg once daily, taken as oral capsules
  Other Names: LENVIMA®; MK-7902; E7080
  Arms: Lenvatinib + Pembrolizumab
Biological: Pembrolizumab — 200 mg 30-minute IV infusion on day 1 of each 21-day cycle
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
  Arms: Lenvatinib + Pembrolizumab
Drug: Docetaxel — 75 mg/m^2 administered as an IV infusion on day 1 of each 21-day cycle
  Other Names: TAXOTERE®
  Arms: SOC Chemotherapy
Drug: Capecitabine — 1250 mg/m^2 twice daily on days 1-14 of each 21-day cycle, taken as oral tablets
  Other Names: Xeloda®
  Arms: SOC Chemotherapy
Drug: Paclitaxel — 80 mg/m^2 administered as an IV infusion on days 1, 8, and 15 of each 21-day cycle
  Other Names: Taxol
  Arms: SOC Chemotherapy
Drug: Cetuximab — 400 mg/m^2 loading dose, followed by 250 mg/m^2 administered as an IV infusion on days 1, 8, and 15 of each 21-day cycle
  Other Names: ERBITUX®
  Arms: SOC Chemotherapy
Drug: Lenvatinib — 24 mg once daily, taken as oral capsules
  Other Names: LENVIMA®; MK-7902; E7080
  Arms: Lenvatinib Monotherapy

SUMMARY:
Researchers are looking for new ways to treat people with head and neck cancer whose cancer has come back after treatment (recurrent) or whose cancer has spread to other parts of the body (metastatic). Some people with recurrent or metastatic head and neck cancer are treated with chemotherapy and immunotherapy, but the cancer gets worse.

The goal of this study is to learn if more people who receive lenvatinib and pembrolizumab have a better overall survival rate than people who receive standard chemotherapy treatment.

DETAILED DESCRIPTION:
With Amendment 7, participants will discontinue lenvatinib and pembrolizumab and lenvatinib monotherapy, unless discussed with the Sponsor.

A protocol-specified periodic safety review was completed with a data cut-off of 31-May-2024 (Primary Completion Date) and served as the final analysis of the primary outcome measure. Per protocol, 34 participants enrolled after the primary completion date and will be analyzed in the End of Trial analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed recurrent (not amenable to curative treatment with local and/or systemic therapies) or metastatic (disseminated) head and neck squamous cell carcinoma (HNSCC) of the oral cavity, oropharynx, hypopharynx, and/or larynx that is considered incurable by local therapies
* Disease progression at any time during or after treatment with a platinum-containing (e.g., carboplatin or cisplatin) regimen
* Disease progression on or after treatment with a programmed cell death protein 1/programmed death-ligand 1 monoclonal antibody (anti-PD-1/PD-L1 mAb)
* Pre-study imaging that demonstrates evidence of disease progression based on investigator review of at least 2 pre-study images per RECIST 1.1, following initiation of treatment with a PD-1/PD-L1 inhibitor
* Measurable disease by computed tomography scan (CT) or magnetic resonance imaging (MRI) based on Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as verified by blinded independent central review (BICR). Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of the first dose of study intervention
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 1 week after the last dose of lenvatinib, 3 months after the last dose of capecitabine and paclitaxel, and 6 months after the last dose of docetaxel:

  * Refrain from donating sperm
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception unless confirmed to be azoospermic
  * Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP)
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 120 days post pembrolizumab or 1 month post lenvatinib, whichever occurs last (Arms 1 and 3), or during the intervention period and for at least 6 months after the last dose of capecitabine, docetaxel, paclitaxel; and 2 months after the last dose of cetuximab (Arm 2)
  * Female participants who randomize to Arm 2 must also agree not to donate or freeze/store eggs during the intervention period and for at least 6 months after the last dose of capecitabine, docetaxel, paclitaxel; and 2 months after the last dose of cetuximab
* Adequately controlled blood pressure (BP) with or without antihypertensive medications
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Adequate organ function

Exclusion Criteria:

* Disease that is suitable for local therapy administered with curative intent
* Life expectancy of less than 3 months and/or has rapidly progressing disease in the opinion of the treating investigator
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids, or has current pneumonitis/interstitial lung disease
* Active infection requiring systemic therapy
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Known additional malignancy that is progressing or has required active systemic treatment within the past 3 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ that have undergone potentially curative therapy
* Active autoimmune disease that has required systemic treatment in the past 2 years
* Had an allogeneic tissue/solid organ transplant
* Known history of human immunodeficiency virus (HIV) infection
* History of any contraindication or has a severe hypersensitivity to any components of pembrolizumab, lenvatinib or SOC chemotherapy.
* Pre-existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
* History of a gastrointestinal malabsorption or any other condition or procedure that may affect oral study drug absorption
* Had major surgery within 3 weeks prior to first dose of study interventions
* Clinically significant cardiovascular impairment within 12 months of the first dose of study drug
* Active tuberculosis
* Has difficulty swallowing capsules or ingesting a suspension orally, or by a feeding tube
* Prior treatment with lenvatinib
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Study Day 1 or has not recovered from adverse events (AEs) due to a previously administered agent. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible
* Has received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention. Note: Administration of killed vaccines is allowed
* Previously treated with 4 or more systemic regimens given for recurrent/metastatic disease
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (120):
- United States (55):
  - City of Hope ( Site 1519), Duarte, California
  - UCLA Hematology/Oncology - Westwood (Building 100) ( Site 1568), Los Angeles, California
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 1505), New Haven, Connecticut
  - Georgetown University Medical Center ( Site 1520), Washington D.C., District of Columbia
  - UF Health ( Site 1554), Gainesville, Florida
  - Mid Florida Hematology and Oncology Center ( Site 1606), Orange City, Florida
  - Cleveland Clinic Florida ( Site 1596), Weston, Florida
  - Georgia Cancer Center at Augusta University ( Site 1575), Augusta, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 1521), Marietta, Georgia
  - Memorial Health University Medical Center ( Site 1626), Savannah, Georgia
  - Beacon Cancer Care ( Site 1599), Post Falls, Idaho
  - Rush University Medical Center ( Site 1560), Chicago, Illinois
  - NorthShore University HealthSystem - Evanston Hospital ( Site 1614), Evanston, Illinois
  - IU Health Ball Memorial Hospital, Inc.-IU Health Ball Memorial Cancer Center ( Site 1612), Muncie, Indiana
  - University of Iowa ( Site 1572), Iowa City, Iowa
  - University of Kansas Cancer Center ( Site 1538), Westwood, Kansas
  - Norton Hospital-Norton Cancer Institute - Downtown ( Site 1601), Louisville, Kentucky
  - Mercy Health-Paducah Cancer Center ( Site 1623), Paducah, Kentucky
  - Our Lady of the Lake RMC-Clinical Research ( Site 1624), Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center Baton Rouge ( Site 1622), Baton Rouge, Louisiana
  - University of Maryland Greenebaum Cancer Center ( Site 1522), Baltimore, Maryland
  - Boston Medical Center ( Site 1605), Boston, Massachusetts
  - University of Massachusetts Chan Medical School ( Site 1616), Worcester, Massachusetts
  - VA Ann Arbor Healthcare System ( Site 1584), Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute ( Site 1566), Detroit, Michigan
  - Henry Ford Health System ( Site 1544), Detroit, Michigan
  - Hattiesburg Clinic ( Site 1515), Hattiesburg, Mississippi
  - Jackson Oncology Associates, PLLC-Clinical Trials ( Site 1625), Jackson, Mississippi
  - Washington University School of Medicine ( Site 1500), St Louis, Missouri
  - St. Vincent Frontier Cancer Center ( Site 1507), Billings, Montana
  - University Of Nebraska Medical Center ( Site 1570), Omaha, Nebraska
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists ( Site 1627), Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 1555), Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 1523), New Brunswick, New Jersey
  - Perlmutter Cancer Center at Winthrop Oncology Hematology Associates NYU Langone Health ( Site 1597), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 1582), New York, New York
  - Levine Cancer Institute ( Site 1590), Charlotte, North Carolina
  - Duke Cancer Institute ( Site 1541), Durham, North Carolina
  - University of Cincinnati Medical Center ( Site 1567), Cincinnati, Ohio
  - University Hospital Cleveland ( Site 1578), Cleveland, Ohio
  - Cleveland Clinic Main ( Site 1598), Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C ( Site 1558), Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 1508), Tulsa, Oklahoma
  - Gettysburg Cancer Center ( Site 1594), Gettysburg, Pennsylvania
  - Penn State Hershey Medical Center ( Site 1561), Hershey, Pennsylvania
  - Fox Chase Cancer Center ( Site 1502), Philadelphia, Pennsylvania
  - Medical University of South Carolina ( Site 1579), Charleston, South Carolina
  - St Francis Cancer Center-Research Office ( Site 1607), Greenville, South Carolina
  - The Center For Cancer And Blood Disorders ( Site 1569), Fort Worth, Texas
  - Utah Cancer Specialists ( Site 1621), Salt Lake City, Utah
  - Huntsman Cancer Institute ( Site 1532), Salt Lake City, Utah
  - Inova Schar Cancer Institute ( Site 1550), Fairfax, Virginia
  - Hematology Oncology Associates of Fredericksburg ( Site 1537), Fredericksburg, Virginia
  - MultiCare Health System-MultiCare Oncology - Puget Sound ( Site 1609), Tacoma, Washington
  - Medical College of Wisconsin Clinical Cancer Center ( Site 1574), Milwaukee, Wisconsin
- Australia (6):
  - Mid North Coast Cancer Institute ( Site 0109), Port Macquarie, New South Wales
  - Blacktown Hospital ( Site 0101), Sydney, New South Wales
  - The Townsville Hospital ( Site 0107), Douglas, Queensland
  - Gallipoli Medical Research Ltd-GMRF CTU ( Site 0105), Greenslopes, Queensland
  - Royal Adelaide Hospital ( Site 0110), Adelaide, South Australia
  - Monash Health ( Site 0102), Clayton, Victoria
- Brazil (2):
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0806), Porto Alegre, Rio Grande do Sul
  - A. C. Camargo Cancer Center ( Site 0809), São Paulo
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 0304), Calgary, Alberta
  - BC Cancer-Vancouver Center ( Site 0306), Vancouver, British Columbia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0307), Hamilton, Ontario
  - Sunnybrook Research Institute ( Site 0308), Toronto, Ontario
- Colombia (4):
  - Instituto de Cancerología ( Site 0408), Medellín, Antioquia
  - Sociedad De Oncologia Y Hematologia Del Cesar ( Site 0404), Valledupar, Cesar Department
  - Administradora Country S.A.S - Clínica del Country ( Site 0407), Bogotá, Cundinamarca
  - IMAT S.A.S ( Site 0409), Montería, Departamento de Córdoba
- Rigshospitalet University Hospital Copenhagen ( Site 1000), Copenhagen, Capital Region, Denmark
- France (6):
  - Hopital La Timone ( Site 0503), Marseille, Bouches-du-Rhone
  - Centre de Cancerologie du Grand Montpellier ( Site 0508), Montpellier, Herault
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne-ONCOLOGY ( Site 0510), Clermont-Ferrand, Puy-de-Dome
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen ( Site 0509), Rouen, Seine-Maritime
  - Institut Gustave Roussy ( Site 0505), Villejuif, Val-de-Marne
  - Institut Curie ( Site 0500), Paris
- Israel (4):
  - Soroka Medical Center-Oncology ( Site 0604), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0602), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0601), Jerusalem
  - Chaim Sheba Medical Center ( Site 0600), Ramat Gan
- Oslo universitetssykehus, Radiumhospitalet ( Site 1102), Oslo, Norway
- Portugal (2):
  - Unidade Local de Saude Gaia/Espinho - Hospital Eduardo Santos Silva ( Site 1401), Vila Nova de Gaia, Porto District
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 1400), Porto
- Romania (7):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L. ( Site 1703), Bucharest, București
  - Spitalul Clinic Colțea ( Site 1708), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 1701), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 1702), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 1706), Floreşti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 1704), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 1707), Timișoara, Timiș County
- South Korea (4):
  - Seoul National University Bundang Hospital ( Site 1801), Seongnam, Kyonggi-do
  - Ajou University Hospital ( Site 1802), Suwon, Kyonggi-do
  - Severance Hospital Yonsei University Health System ( Site 1800), Seoul
  - Samsung Medical Center ( Site 1803), Seoul
- Spain (7):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 0700), L'Hospitalet de Llobregat, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA ( Site 0707), Barcelona, Catalonia
  - Centro Oncologico de Galicia ( Site 0706), A Coruña, Galicia
  - Hospital General de Valencia ( Site 0703), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d Hebron ( Site 0701), Barcelona
  - Hospital Ramon y Cajal ( Site 0705), Madrid
  - Hospital Virgen de la Victoria ( Site 0702), Málaga
- Taiwan (7):
  - Chang Gung Medical Foundation - Kaohsiung ( Site 1204), Kaohsiung City
  - China Medical University Hospital ( Site 1205), Taichung
  - Taichung Veterans General Hospital ( Site 1206), Taichung
  - National Cheng Kung University Hospital ( Site 1202), Tainan
  - National Taiwan University Hospital ( Site 1200), Taipei
  - Taipei Veterans General Hospital ( Site 1201), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 1203), Taoyuan District
- United Kingdom (10):
  - Aberdeen Royal Infirmary ( Site 0911), Aberdeen, Aberdeen City
  - Castle Hill Hospital ( Site 0910), Cottingham, East Riding Of Yorkshire
  - The Beatson West of Scotland Cancer Centre ( Site 0909), Glasgow, Glasgow City
  - Guy s and St Thomas Hospital NHS Foundation Trust ( Site 0903), London, Great Britain
  - University Hospital Southampton NHS Foundation Trust ( Site 0905), Southampton, Hampshire
  - Royal Marsden Hospital ( Site 0902), London, London, City of
  - Charing Cross Hospital ( Site 0908), London, London, City of
  - Musgrove Park Hospital ( Site 0904), Taunton, Somerset
  - Royal Marsden Hospital. ( Site 0901), Sutton, Surrey
  - The Christie NHS Foundation Trust ( Site 0907), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Taylor MH, Schmidt EV, Dutcus C, Pinheiro EM, Funahashi Y, Lubiniecki G, Rasco D. The LEAP program: lenvatinib plus pembrolizumab for the treatment of advanced solid tumors. Future Oncol. 2021 Feb;17(6):637-648. doi: 10.2217/fon-2020-0937. Epub 2020 Dec 10. PMID 33300372
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26315&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol-specified final analysis for the results, including participant flow, was performed on 374 participants enrolled within the primary completion data cut-off. Analysis of the remaining 34 participants will be included in the End of Trial analysis.
  Participants who experienced progressive disease in the lenvatinib monotherapy or Standard of Care arms could switch over to receive lenvatinib + pembrolizumab. One participant switched over and received only pembrolizumab.
Groups:
- Lenvatinib + Pembrolizumab: Participants were treated with the combination of lenvatinib (once daily 20 mg oral dose) plus pembrolizumab (200 mg 30-minute intravenous (IV) infusion on Day 1 of each 21-day cycle for 35 cycles), until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
- SOC Chemotherapy: Participants were treated with investigator's choice of standard of care (SOC) chemotherapy (docetaxel, paclitaxel, cetuximab, or capecitabine) until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
- Lenvatinib Monotherapy: Participants were treated with lenvatinib monotherapy (once daily 24 mg oral dose) until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy
Started | 144 | 142 | 88
Treated | 143 | 140 | 88
Switched Over to Pembrolizumab + Lenvatinib | 0 | 61 | 18
Switched Over to Pembrolizumab | 0 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 144 | 142 | 88
Not completed — Death | 100 | 86 | 57
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Participant Ongoing in Study | 41 | 53 | 28

BASELINE CHARACTERISTICS:
Population: Per protocol, analysis population consisted of all participants randomized by the primary completion data cut-off.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy | Total
Number analyzed (Participants) | 144 | 142 | 88 | 374
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (9.0) | 61.4 (10.0) | 59.9 (9.3) | 61.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 14 | 51
  Male | 126 | 123 | 74 | 323
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6 | 12
  Not Hispanic or Latino | 139 | 137 | 82 | 358
  Unknown or Not Reported | 2 | 2 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3 | 6
  Asian | 35 | 40 | 25 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 8
  White | 104 | 96 | 57 | 257
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG = 0 | 52 | 58 | 32 | 142
    ECOG = 1 | 92 | 84 | 56 | 232
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (<50% or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS = <50% | 121 | 120 | 74 | 315
    TPS = ≥ 50% | 23 | 22 | 14 | 59

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to approximately 45 months
Population: The analysis population consisted of all participants who were randomized prior to the primary completion data cut-off. Per protocol, participants who received lenvatinib monotherapy were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy
Number analyzed (Participants) | 144 | 142 | 0
Months | 8.4 [6.9 to 10.3] | 11.3 [9.8 to 14.4] |
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs SOC Chemotherapy; Test type: Superiority; p = 0.9963, Log Rank — One-sided p-value based on log-rank test stratified by baseline PD-L1 TPS (<50% versus ≥50%) and baseline ECOG performance status (0 versus 1). The reported p-value is nominal; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [1.11 to 1.97] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by baseline PD-L1 TPS (<50% versus ≥50%) and baseline ECOG performance status (0 versus 1)

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Responses were according to modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by blinded independent central review (BICR). RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD.
Time Frame: Up to approximately 45 months
Population: The analysis population consisted of all participants randomized by the primary completion data cut-off. Per protocol, participants who received lenvatinib monotherapy were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy
Number analyzed (Participants) | 144 | 142 | 0
Months | 3.0 [2.8 to 3.9] | 2.8 [2.6 to 4.0] |
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs SOC Chemotherapy; Test type: Superiority; p = 0.4181, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.74 to 1.28] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of the diameters of target lesions) until progressive disease (PD) or death due to any cause, whichever occurred first. Responses were according to modified RECIST 1.1 as assessed by BICR. RECIST 1.1 was modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to approximately 45 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy
Number analyzed (Participants) | 144 | 142 | 0
Percentage of Participants | 13.9 [8.7 to 20.6] | 20.4 [14.1 to 28.0] |
Statistical Analysis 1: Comparison: Lenvatinib + Pembrolizumab vs SOC Chemotherapy; Test type: Superiority; p = 0.9266219, Miettinen & Nurminen; One-sided p-value for testing H0: difference in % = 0 versus H1: difference in % > 0. The reported p-value is nominal; Difference in Percentage = -6.5, 95% CI 2-sided [-15.4 to 2.3] — Based on Miettinen & Nurminen method stratified by baseline PD-L1 TPS (<50% versus ≥50%) and baseline ECOG performance status (0 versus 1)

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented evidence of complete response (CR: disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of the diameters of target lesions) until progressive disease (PD) or death due to any cause, whichever occurred first. Responses were according to modified RECIST 1.1 as assessed by BICR.
Time Frame: Up to approximately 45 months
Population: The analysis population consisted of all participants randomized by the primary completion data cut-off who experienced a confirmed CR or PR. Per protocol, participants who received lenvatinib monotherapy were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy
Number analyzed (Participants) | 20 | 29 | 0
Months | 4.1 [3.6 to 7.9] | 5.9 [3.7 to 11.8] |

5. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE was presented.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE was presented.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 45 months
Description: Serious & Other AEs includes participants randomized by primary completion data cut-off who received ≥1 dose of study drug. All-Cause Mortality includes participants randomized by primary completion data cut-off. Per protocol, progression of cancer was not considered an AE unless related to study treatment. MedDRA terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. AEs are reported by treatment received.
Groups:
- SOC Chemotherapy Switched Over to Pembrolizumab+Lenvatinib: Participants who experienced centrally verified progressive disease (PD) on SOC chemotherapy switched over with Sponsor consultation and received a combination of lenvatinib (once daily 20 mg oral dose) plus pembrolizumab (200 mg 30-minute IV infusion on Day 1 of each 21-day cycle for up to 35 cycles) until a protocol-specified discontinuation criterion was met.
- SOC Chemotherapy Switched Over to Pembrolizumab: Participants who experienced centrally verified progressive disease (PD) on SOC chemotherapy switched over with Sponsor consultation and received pembrolizumab (200 mg 30-minute IV infusion on Day 1 of each 21-day cycle for up to 35 cycles) until a protocol-specified discontinuation criterion was met.
- Lenvatinib Switched Over to Pembrolizumab+Lenvatinib: Participants who experienced centrally verified progressive disease (PD) on lenvatinib monotherapy switched over with Sponsor consultation and received a combination of lenvatinib (once daily 20 mg oral dose) plus pembrolizumab (200 mg 30-minute IV infusion on Day 1 of each 21-day cycle for up to 35 cycles) until a protocol-specified discontinuation criterion was met.
Arm/Group | Lenvatinib + Pembrolizumab | SOC Chemotherapy | Lenvatinib Monotherapy | SOC Chemotherapy Switched Over to Pembrolizumab+Lenvatinib | SOC Chemotherapy Switched Over to Pembrolizumab | Lenvatinib Switched Over to Pembrolizumab+Lenvatinib
All-Cause Mortality (participants affected / at risk) | 103/144 | 42/142 | 50/88 | 44/61 | 1/1 | 10/18
Serious Adverse Events (participants affected / at risk) | 86/143 | 57/140 | 45/88 | 27/61 | 1/1 | 6/18
Other Adverse Events (participants affected / at risk) | 139/143 | 135/140 | 80/88 | 55/61 | 1/1 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=143) | SOC Chemotherapy (N=140) | Lenvatinib Monotherapy (N=88) | SOC Chemotherapy Switched Over to Pembrolizumab+Lenvatinib (N=61) | SOC Chemotherapy Switched Over to Pembrolizumab (N=1) | Lenvatinib Switched Over to Pembrolizumab+Lenvatinib (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 20 (23) | 8 (8) | 4 (4) | 5 (6) | 1 (1) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 2 (2) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 3 (4) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post infection glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper airway necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab (N=143) | SOC Chemotherapy (N=140) | Lenvatinib Monotherapy (N=88) | SOC Chemotherapy Switched Over to Pembrolizumab+Lenvatinib (N=61) | SOC Chemotherapy Switched Over to Pembrolizumab (N=1) | Lenvatinib Switched Over to Pembrolizumab+Lenvatinib (N=18)
Anaemia (Blood and lymphatic system disorders) | 20 (24) | 37 (40) | 13 (18) | 4 (4) | 0 (0) | 2 (2)
Necrotic lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 49 (52) | 12 (12) | 28 (28) | 15 (15) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 4 (4) | 9 (11) | 4 (4) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 7 (9) | 1 (1) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 25 (28) | 32 (38) | 20 (24) | 6 (7) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 38 (48) | 26 (35) | 25 (39) | 15 (20) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 5 (5) | 10 (10) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 5 (6) | 3 (4) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 12 (13) | 9 (10) | 9 (10) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 7 (7) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 26 (30) | 31 (43) | 12 (13) | 12 (14) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 6 (8) | 5 (5) | 6 (6) | 2 (4) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 11 (11) | 3 (3) | 6 (8) | 4 (4) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 52 (73) | 28 (30) | 26 (34) | 21 (26) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 18 (20) | 13 (16) | 10 (10) | 5 (6) | 0 (0) | 2 (2)
Asthenia (General disorders) | 30 (33) | 31 (46) | 23 (26) | 7 (7) | 0 (0) | 3 (4)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 37 (38) | 24 (24) | 20 (23) | 12 (13) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 6 (8) | 9 (9) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 13 (15) | 9 (12) | 5 (7) | 4 (4) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Xerosis (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 10 (11) | 6 (6) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 15 (21) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (9) | 7 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (9) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (12) | 8 (11) | 5 (9) | 2 (2) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 4 (4) | 5 (7) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 13 (14) | 11 (19) | 9 (12) | 6 (12) | 1 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 9 (9) | 3 (6) | 3 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 7 (7) | 5 (6) | 5 (6) | 1 (3) | 0 (0) | 3 (3)
Blood thyroid stimulating hormone increased (Investigations) | 3 (3) | 2 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 6 (8) | 9 (14) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (4) | 24 (42) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 8 (11) | 3 (5) | 9 (14) | 3 (6) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 26 (28) | 22 (24) | 27 (28) | 7 (7) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 34 (35) | 27 (29) | 21 (22) | 12 (13) | 0 (0) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (4) | 4 (5) | 2 (2) | 0 (0) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 9 (11) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (7) | 7 (11) | 2 (4) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (10) | 3 (3) | 6 (7) | 3 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (14) | 8 (8) | 6 (12) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7) | 12 (17) | 6 (10) | 3 (5) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9) | 4 (5) | 9 (10) | 1 (1) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (7) | 6 (6) | 3 (10) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 7 (9) | 12 (16) | 4 (6) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (11) | 6 (6) | 1 (1) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 6 (7) | 3 (3) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 13 (13) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 10 (11) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 8 (9) | 1 (1) | 0 (0) | 2 (2)
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 11 (13) | 8 (9) | 9 (9) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 18 (19) | 15 (15) | 11 (12) | 4 (4) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 11 (16) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 16 (19) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 13 (14) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 24 (32) | 5 (5) | 20 (30) | 11 (12) | 0 (0) | 3 (4)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 21 (22) | 9 (9) | 5 (5) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 2 (2) | 7 (7) | 5 (5) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 18 (18) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 7 (8) | 1 (1) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 4 (7) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 7 (7) | 11 (17) | 3 (3) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 12 (12) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 23 (23) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 22 (24) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 13 (13) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (20) | 7 (11) | 11 (11) | 9 (10) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (11) | 4 (4) | 4 (5) | 2 (2) | 0 (0) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 14 (14) | 26 (31) | 7 (7) | 5 (5) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 60 (77) | 5 (6) | 34 (43) | 17 (19) | 1 (1) | 1 (3)
Hypotension (Vascular disorders) | 10 (12) | 5 (5) | 4 (5) | 2 (3) | 0 (0) | 3 (3)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT04428151/Prot_SAP_000.pdf